CLINICAL TRIAL: NCT02353975
Title: An Open Label, Randomized, Two-period, Crossover Study to Assess the Effect of Food on SHR3824 and Mass Balance Study in Healthy Volunteers
Brief Title: Effect of a High-fat Meal on the Pharmacokinetics of SHR3824 and Mass Balance Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR3824-104
Record Dates: First submitted 2015-01-20; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes
Keywords: SHR3824; food effect; mass; balance; Phase I
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Arachnodactyly | interventions — henagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHR3824 10mg fasted to fed (Experimental): SHR3824 tablet, fasting conditions day 1, visit 2, 7 days wash-out, SHR3824 tablet, high fat, high calorie breakfast day 1, visit 3.
  Interventions: Drug: SHR3824
- SHR3824 10mg fed to fasted (Experimental): SHR3824, high fat, high calorie breakfast day 1, visit 2, 7 days wash-out, SHR3824, fasting conditions day 1, visit 3.
  Interventions: Drug: SHR3824

INTERVENTIONS:
Drug: SHR3824 — SHR3824 tablet,10mg, fasting conditions and high fat, high calorie breakfast.

SUMMARY:
This open-label, randomized, two-period, two-treatment (single doses of 10 mg SHR3824 fasted or fed), crossover study was conducted to evaluate the effect of a high-fat meal on the pharmacokinetics of SHR3824 and mass balance study in 12 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* BMI 18-25 kg/m2.

Exclusion Criteria:

* History of clinically significant illness.
* History of alcohol or drug abuse.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SHR3824 | Day 1-4 on visit 2 and visit 3
  Cmax (a measure of the body's exposure to SHR3824) will be compared under fating state and fasted state
The area under the plasma concentration-time curve (AUC) of SHR3824 | Day 1-4 on visit 2 and visit 3
  AUC (a measure of the body's exposure to SHR3824) will be compared under fating state and fasted state
The accumulative excretion rate of SHR3824 and its metabolites in urine and feces | Day 1-4 on visit 2 and visit 3
  Accumulative excretion rate will be compared under fating state and fasted state

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability. | Up to Day 12